CLINICAL TRIAL: NCT00613353
Title: Sedentary Behavior in Overweight Women
Status: Completed | Type: Observational
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Jacinda Roach, Assistant Professor, Department of Medicine, The University of Mississippi Medical Center
Other Study IDs: 2007-0150; DHHS FWA#00003630
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Sedentary Behavior; Overweight
Keywords: Female
MeSH Terms: conditions — Sedentary Behavior; Overweight

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- I: Caucasian and African American females between the ages of 18 and 65.
  Interventions: Other: Behavioral

INTERVENTIONS:
Other: Behavioral — Participants will be asked to wear an accelerometer

SUMMARY:
Objective activity data will be collected using accelerometry for a minimum of seven days on 38 adult, female, women recruited from the metabolic Clinic at the University of Mississippi Medical Center. Following objective measurement of activity, participants will complete self-report and objective activity data, as well as the relationship between sedentary activities and food cravings will be examined. It is hypothesized that minutes of sedentary behavior, especially time spent in television viewing, will be significantly correlated with total and specific food cravings.

ELIGIBILITY:
Inclusion Criteria: Caucasian or African American women between the ages of 18 and 65

Exclusion Criteria: Males and women who are younger than 18 and older than 65

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caucasian or African American women between the ages of 18 and 65.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Minutes of sedentary behavior, especially time spent in television viewing, will be significantly correlated with total and specific food cravings | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacinda B Roach, PhD, Principal Investigator — The University of Mississippi Medical Center
Locations (1):
- The University of Mississippi Medical Center, Jackson, Mississippi, United States